CLINICAL TRIAL: NCT02149485
Title: Long-term Safety of Preimplantation Genetic Diagnosis. Follow-up of 5-year Old Children Born After PGD.
Brief Title: Follow-up of 5-year Old Children Born After PGD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Christine de Die- Smulders, prof. dr., Maastricht University Medical Center
Other Study IDs: 13-2010
Record Dates: First submitted 2014-05-20; First posted 2014-05-29 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Preimplantation Genetic Diagnosis
Keywords: PGD,; follow up

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Since 1995, preimplantation genetic diagnosis (PGD) has been performed in The Netherlands for couples at high risk for transmitting severe or lethal genetic conditions or who have experienced multiple miscarriages due to chromosomal translocations. Approximately 260 children have been born after PGD in The Netherlands. Follow-up data on children born after PGD are scarce. Long-term studies on PGD children have not been conducted in The Netherlands. Results of studies in other countries on 2-year old PGD children are reassuring. These children and their parents have normal scores on relevant parameters such as general health, cognitive and socioemotional development, parent-child interaction and parental stress. Studies of good methodological quality of older children have not yet been published.

Objective: Long-term follow-up of children who have been born after PGD in The Netherlands. The primary aim is to assess the safety of PGD with regard to the health and development of the children.

Study design: A cohort study. Study population: 5- and 8 year old children born after PGD in The Netherlands for various indications and their parents. Control groups consist of 5 and 8-year old naturally conceived (NC) children of parents who have considered PGD treatment and 5 and 8-year old children born after in vitro fertilisation/intracytoplasmatic sperm injection (IVF/ICSI), and the parents of the two latter groups of children.

DETAILED DESCRIPTION:
Parents are asked to fill out questionnaires on their own and their child's medical history. A physical examination of the children will be performed, a swab for collection of buccal cells for (future) DNA methylation analysis will be taken and their cognitive and socioemotional development will be assessed. In the 8 years old children cardiovascular status will be evaluated.

Main study parameters: general health, cognitive and socioemotional development, parent-child interaction and parental stress.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

The study procedure consists of filling out questionnaires by parents and a one-time visit to the hospital. No invasive interventions will be performed, except 1 tube of blood in the 8 year old group. The risks associated with the study procedure are very small. The results provide more information about the risks of PGD to prospective parents who are considering PGD and to healthcare providers involved in PGD treatment.

ELIGIBILITY:
Inclusion criteria:

PGD children

* 5-year old singleton PGD children with Caucasian parents
* Children must have the Dutch language as their mother tongue for participation in the intelligence quotient (IQ) test. Children that do not have Dutch as their mother tongue will be excluded from the IQ test, but can take part in the rest of the procedure

Naturally conceived (NC) children

* 5-year old singleton NC children with Caucasian parents, matched with PGD children on age and sex
* Parents must have attended the PGD clinic in Maastricht for an informative consultation
* Parents must have become pregnant without any assisted reproductive technique
* Children must have the Dutch language as their mother tongue

IVF/ICSI children

* 5-year old singleton IVF/ICSI children with Caucasian parents, matched with PGD children on age and sex
* Children must have the Dutch language as their mother tongue

Exclusion criteria:

PGD children

* Twins or triplets
* Parents of non-Caucasian descent
* Children with known chromosomal abnormalities (e.g. trisomy 21) or gene disorders with childhood expression of symptoms

NC children

* Twins or triplets
* Parents of non-Caucasian descent
* Children with known chromosomal abnormalities or gene disorders with childhood expression of symptoms

IVF/ICSI children

* Twins or triplets
* Parents of non-Caucasian descent
* Children with known chromosomal abnormalities or gene disorders with childhood expression of symptoms

  8 years old group Former participants of the study in 5 year old children

Ages: 5 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 5 years old children born after preimplantation genetic diagnosis
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Physical health of 5 years old children born after preimplantation genetic diagnosis | 5 years
  Physical health of 5 and 8 years old children born after PGD will be assessed by physical examination and measurement of height, weight and compared with children born after IVF/ICSI and naturally conceived children.

SECONDARY OUTCOMES:
Psychological health of 5 and 8 years old children born after preimplantation genetic diagnosis | 5 years
  Psychological health will be assesses by neuropsychological testing, and questionaires

CONTACTS AND LOCATIONS:
Overall Officials: Christine de Die-Smulders, MD PhD, Principal Investigator — Maastricht University Hospital
Locations (2):
- Netherlands (2):
  - Maastricht University Hospital, Maastricht, Limburg
  - University Medical Center Utrecht, Utrecht, Utrecht

REFERENCES:
- [Derived] Heijligers M, Peeters A, van Montfoort A, Nijsten J, Janssen E, Gunnewiek FK, de Rooy R, van Golde R, Coonen E, Meijer-Hoogeveen M, Broekmans F, van der Hoeven M, Arens Y, de Die-Smulders C. Growth, health, and motor development of 5-year-old children born after preimplantation genetic diagnosis. Fertil Steril. 2019 Jun;111(6):1151-1158. doi: 10.1016/j.fertnstert.2019.01.035. Epub 2019 Apr 17. PMID 31005312
- [Derived] Heijligers M, Verheijden LMM, Jonkman LM, van der Sangen M, Meijer-Hoogeveen M, Arens Y, van der Hoeven MA, de Die-Smulders CEM. The cognitive and socio-emotional development of 5-year-old children born after PGD. Hum Reprod. 2018 Nov 1;33(11):2150-2157. doi: 10.1093/humrep/dey302. PMID 30265304